CLINICAL TRIAL: NCT05928871
Title: The Effect of Pre-operative Versus Post-operative Misoprostol in Reducing Blood Loss During and After Elective Cesarean Section.
Brief Title: Pre Versus Post-operative Misoprostol in Reducing Blood Loss After Cesarean Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AN2023-2
Record Dates: First submitted 2023-06-24; First posted 2023-07-03 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Misoprostol Allergy
Keywords: misoprostol; cesarean section; postpartum hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preop (Active Comparator): 60 women: will receive preoperative 600 microgram of misoprostol ( 3 tablets ) rectally after spinal anaesthesia and urinary catheterization and postoperative placebo (3 tablets). (as per WHO dose recommendation)
  Interventions: Drug: Misoprostol 200mcg Tab
- postop (Active Comparator): 60 women: will receive preoperative placebo "3 tablets" and postoperative 600 microgram of misoprostol " 3 tablets" at operating theatre (as per WHO dose recommendation).
  Interventions: Drug: Misoprostol Pill

INTERVENTIONS:
Drug: Misoprostol 200mcg Tab — 60 women: will receive preoperative 600 microgram of misoprostol ( 3 tablets ) rectally after spinal anaesthesia and urinary catheterization and postoperative placebo (3 tablets). (as per WHO dose recommendation)
  Other Names: Misotac
  Arms: preop
Drug: Misoprostol Pill — 60 women: will receive preoperative placebo "3 tablets" and postoperative 600 microgram of misoprostol " 3 tablets" at operating theatre (as per WHO dose recommendation).
  Other Names: misotac
  Arms: postop

SUMMARY:
Cesarean section is the most common performed major surgical interventions among women all over the world.Cesarean section has many serious complications, including primary postpartum hemorrhage (PPH). Postpartum hemorrhage is one of the most serious causes of maternal mortality and morbidity, especially in developing countries, and the number of maternal deaths due to postpartum hemorrhage is estimated to exceed 100,000 maternal deaths each year. The incidence of CS is increasing and the average blood loss during CS (1000 mL) is double the amount lost during vaginal delivery (500 mL) .

The most successful technique for decreasing PPH is active management of the third stage of labor (AMTSL), requires prophylactic utero-tonic drugs as oxytocin, ergometrine malate and combinations of them , They must be administered by injection.

Misoprostol is synthetic prostaglandin (PGE1 analogue), with utero-tonic properties, has been proposed as an alternative strategy for prevention of PPH in settings where oxytocin use is not handy. It has important advantages over oxytocin, including the potential for oral administration and a long shelf life at room temperature.Misoprostol is affordable and widely available, can be easily administered via multiple routes, and has a good safety profile if properly administered and monitored, all of which makes it an alternative treatment option of PPH in developing countries.

Investigators were comparing the effect of preoperative and post-operative rectally administrated misoprostol on operative blood loss at cesarean section. Misoprostol has an important effect in terms of decreased postoperative morbidity and a decrease in risks associated with blood transfusions.

DETAILED DESCRIPTION:
History taking:

* Verbal consent.
* Detailed clinical history.
* Personal history:

Name, Age, Parity, Occupation, Residency and Special habits.

- Present history: History of onset, course and duration of vaginal bleeding or bloody vaginal discharge, presence of uterine contraction, PROM, IUGR or any indication for cesarean section.

- Obstetric history: History of previous preterm labor, previous abortion, previous full term deliveries, RH incompatibility, mode of delivery and fetal outcome.

- Menstrual history: For estimation of gestational age using Naegele's rule, provided that she had regular cycles for the last three months before she got pregnant and was not taking contraceptive pills during this period and she was sure of her dates.

Term pregnancy defined as delivery between 37 and 42 weeks of gestation. Gestational age was assessed from the menstrual history and confirmed by measurement of fetal crown-rump length at a first-trimester scan.

- Past history: History of medical disorders, drug therapy or allergy or history of intake of other tocolytic drugs.

- Family history : For any similar condition

Examination

* Full clinical examination (pulse, temperature and the blood pressure).
* General examination including blood pressure, heart rate, body temperature, body mass index, head& neck examination, Bilateral lower limb examination, chest, heart and abdominal examination for fundal level.
* Local clinical examination; assessment of maternal health, obstetric abdominal examination for: fundal level, fetal presentation, estimating fetal weight and scars of previous operations, uterine contraction if present, auscultation of FHR. Vaginal examination will be done to detect condition of cervix (dilatation and effacement).
* Routine antenatal investigations (Rh, CBC, HTC, Hb, Coagulation profile, fasting and postprandial blood sugar and complete urine analysis).
* Ultrasonography examination : to assess the following data:
* Gestational age
* Fetal viability
* Fetal presentation and EFW.
* Exclusion of any fetal congenital anomalies.
* To ensure that the all inclusion criteria are present.
* Check amniotic fluid index.

Intervention:

Cesarean section will be done by a senior registrar who performed at least 300 cesarean sections before the start of the study.

All CS will be performed using spinal anesthesia, the abdomen is entered by Pfannenstiel abdominal incision. After induction of anesthesia,patients assigned to group 1 will receive rectal misoprostol immediately after urinary catheterization and before skin incision. Participants are assigned to group 2 will receive 600μg rectal misoprostol immediately after skin closure. all women will be received 5IU of oxytocin by slow intravenous after cord clamping (British Medical, Royal Pharmaceutical society of Great British, 2011).

Sterilization and toweling of the patient then the standard technique of trans-peritoneal lower segment cesarean will be adopted.The placenta will be removed by cord traction and uterinecompression. The uterus will be exteriorized and compressed duringclosure which will be achieved by continuous unlocked sutures in 2 layers using Ethicon Vicryl 0 suture. The peritoneum and muscle is closed by Vicryl 0 suture and The sheath is closed by Vicryl 1, and the skin is closed by subcutical suture using proline double zero suture in both groups. Estimation of blood loss was started after skin incision.

* The linen towels will be weighted in (mg) with its cover before and after the operation using a highly accurate digital balance and the difference in weight between dry and soaked linen towels will be calculated.
* Blood loss during the operation will be calculated as follows:
* Volume of the contents of the suction bottle (ml) (A).
* Difference in weight of linen towels (gm) (B) (weight of soaked linen towels (gm) - weight of dry linen towels (gm)).
* Amniotic fluid volume (ml) (C).
* So blood loss during operation (ml) = (A + B) - C (Lapaire et al., 2006).
* Allowable blood loss was calculated for all women according to the underlying law .

ABL= EBV x (Hi - Hf) Hi Hi = initial Hct Hf = final lowest acceptable Hct Estimated Blood Volume (EBV) EBV = weight (kg) X average blood volume (65-75 ml/kg )

* A trained nurse will be responsible for collection of wound dressing placed in vulval area during the first 24 hours after surgery and the difference in weight will be calculated. The overall blood loss will be calculated.
* Changes in hemoglobin concentration and hematocrit value will be measured 24 hours after the cesarean section.
* The need for additional utero-tonic drugs will be given according to the attendant consultant decision or a blood loss more than 1000ml intra operative.
* Operative time, need for blood transfusion and side effects of study drug e.g. nausea, vomiting, diarrhea will be recorded.
* All the patients will receive non-steroidal anti-inflammatory preparation in the form of (Rheumarene®) 75mg IM (one ampoule) immediately postoperative then one ampoule 12 hours postoperative and the need for extra analgesics will be recorded & the degree of postoperative pain will be estimated using visual analogue scale will be done (3 hours and 24 hours) after the operation.
* The Apgar score of the fetus at 1 and 5 minutes, the need for neonatal intensive care unit (NICU) admission and neonatal death will be assessed in the two groups.
* Data were collected and tabulated and statistically analyzed by IBM computer using the Statistical Package for the Social Sciences (SPSS version 15). Chi-square test was used to compare qualitative variables between groups and Fisher exact test was used instead of Chisquare test when the expected cell count is less than 5. Student t-test was used to compare the quantitative variables in parametricdata. p value <0.05 was set signiﬁcant.

ELIGIBILITY:
Inclusion Criteria:

* Women booked for elective cesarean section not in active labor
* Scheduled for primary elective caesarian section.
* No contraindications to prostaglandins.
* Have no history of coagulopathy.
* Aged between 18-40 years.
* Full term pregnancies (GA 37 to 42 weeks).
* Singleton pregnancies.
* BMI 20-30 kg/ m2

Exclusion Criteria:

* Placenta previa.
* Maternal hypertension and Pre-eclampsia. .
* Diabetes mellitus.
* Previous CS and those with active labor.
* Multiple Fibroid uterus .
* Multiple pregnancies.
* Overdistended uterus eg. polyhydramnios
* Previous myomectomy, previous history of PPH .
* Contraindication to spinal anesthesia.
* Blood coagulopathy and bleeding disorder.
* Marked maternal anemia (Preoperative hemoglobin <9 gm/dl).
* Contraindications to prostaglandin therapy (e.g. history of severe bronchial asthma or allergy to misoprostol.
* Extreme of BMI (<20 or >30Kg/m2).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients will be recruited in this study those attending labor ward at kasr el ainy hospital for elective cesarean section
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Estimation of Intraoperative and postoperative blood loss. | 24 hours
  calculate total blood loss in guaze and suction bottle

SECONDARY OUTCOMES:
Need of extra utero-tonic drugs | 24 hours
  use of more uterotonic drugs as oxytocin and ergometrin
Incidence of postpartum hemorrhage. | 24 hours
  blood loss more than 1000 ml
The incidence of side effects e.g. nausea, vomiting, diarrhea, shivering and headache. | 24 hours
  occurance of side effect within 24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Taymour, MD, Principal Investigator — Cairo University
Locations (1):
- faculty of medicine, Kasr el ainy hospital, Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mousa H, Alfirevic Z. (2009): Treatment for primary postpartum hemorrhage (Cochrane review). Chichcster (UK): John Wiley&Sons Ltd. The Cochrane Library; Issue4
- [Background] Tang OS, Schweer H, Seyberth HW, Lee SW, Ho PC. Pharmacokinetics of different routes of administration of misoprostol. Hum Reprod. 2002 Feb;17(2):332-6. doi: 10.1093/humrep/17.2.332. PMID 11821273
- [Result] Is the time of administration of misoprostol of value? The uterotonic effect of misoprostol given pre-and post-operative after elective cesarean section. Middle East Fertility Society Journal, 19(1), 8-12.
- [Result] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin: Clinical Management Guidelines for Obstetrician-Gynecologists Number 76, October 2006: postpartum hemorrhage. Obstet Gynecol. 2006 Oct;108(4):1039-47. doi: 10.1097/00006250-200610000-00046. PMID 17012482
- [Result] Cunningham F. G., Leveno K. J., Bloom Steven L., Hauth John C., Dwight J. Rouse, Dwight J. Rouse. (2001): William's Obstetrics 23rd Edition ISBN: 0071497013, ISBN-13: 9780071497015, PUB. PUBLISHER: The McGraw-Hill Companies.
- [Result] British Medical Association, Royal Pharmaceutical Society of Great Britain (2011): British National Formulary. Cesarean section: an entire guideline. 2011. London.
- [Result] Derman RJ, Kodkany BS, Goudar SS, Geller SE, Naik VA, Bellad MB, Patted SS, Patel A, Edlavitch SA, Hartwell T, Chakraborty H, Moss N. Oral misoprostol in preventing postpartum haemorrhage in resource-poor communities: a randomised controlled trial. Lancet. 2006 Oct 7;368(9543):1248-53. doi: 10.1016/S0140-6736(06)69522-6. PMID 17027730
- [Result] Khan RU, El-Refaey H. Pharmacokinetics and adverse-effect profile of rectally administered misoprostol in the third stage of labor. Obstet Gynecol. 2003 May;101(5 Pt 1):968-74. doi: 10.1016/s0029-7844(03)00174-1. PMID 12738159
- [Result] Langenbach C. Misoprostol in preventing postpartum hemorrhage: a meta-analysis. Int J Gynaecol Obstet. 2006 Jan;92(1):10-8. doi: 10.1016/j.ijgo.2005.10.001. Epub 2005 Nov 23. PMID 16309682
- [Result] Lapaire O, Schneider MC, Stotz M, Surbek DV, Holzgreve W, Hoesli IM. Oral misoprostol vs. intravenous oxytocin in reducing blood loss after emergency cesarean delivery. Int J Gynaecol Obstet. 2006 Oct;95(1):2-7. doi: 10.1016/j.ijgo.2006.05.031. Epub 2006 Aug 23. PMID 16934269
- [Result] Magann EF, Evans S, Hutchinson M, Collins R, Lanneau G, Morrison JC. Postpartum hemorrhage after cesarean delivery: an analysis of risk factors. South Med J. 2005 Jul;98(7):681-5. doi: 10.1097/01.SMJ.0000163309.53317.B8. PMID 16108235
- [Result] Mathai M, Hofmeyr GJ, Mathai NE. Abdominal surgical incisions for caesarean section. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD004453. doi: 10.1002/14651858.CD004453.pub3. PMID 23728648